CLINICAL TRIAL: NCT02795494
Title: Validation and Reliability Testing of the Western Ontario and McMaster Osteoarthritis Scale (WOMAC) Hip Score in Children and Adolescents With Perthes Disease
Brief Title: WOMAC Hip Score in Children and Adolescents With Perthes Disease
Acronym: WOMAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Pediatric Orthopaedic Surgeon, British Columbia Children's Hospital
Other Study IDs: H0700752
Record Dates: First submitted 2016-05-26; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Legg-Calvé-Perthes Disease
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Perthes Group: Participants with Perthes disease. Will be given WOMAC questionnaire at baseline and WOMAC questionnaire at 2 weeks, and ASK-P questionnaire at baseline.
  Interventions: Behavioral: WOMAC questionnaire at baseline; Behavioral: ASK-P questionnaire at baseline; Behavioral: WOMAC questionnaire at 2 weeks
- Fracture Control Group: Participants with an upper extremity fracture but no hip-related conditions. Will be given WOMAC questionnaire at baseline.
  Interventions: Behavioral: WOMAC questionnaire at baseline

INTERVENTIONS:
Behavioral: WOMAC questionnaire at baseline — Patient-reported pain, stiffness and physical function outcome score
Behavioral: ASK-P questionnaire at baseline — Patient-reported activity level score
  Groups: Perthes Group
Behavioral: WOMAC questionnaire at 2 weeks — Patient-reported pain, stiffness and physical function outcome score
  Groups: Perthes Group

SUMMARY:
Patient oriented clinical outcomes have increased in use and popularity and provide a comprehensive assessment of the level of symptoms and function experienced by a patient. Though several measures have been developed and shown to be valid, reliable, and responsive in adults, such efforts have only been rarely undertaken in pediatric populations. Specifically, there has been no validation of the predominant adult hip specific outcome measures, such as the WOMAC and Oxford-12, in children and adolescents. Prior to using such measures in pediatric patients, it is necessary to establish the psychometric properties of these measurements in this population.

The objective of this study is to determine the reliability and validity of the WOMAC hip scores in a pediatric population, between five and nineteen years of age, with Perthes disease. The results of this study will accomplish the above goal, thereby allowing either for widespread use of these measures in pediatric hip disorders or emphasizing the necessity for development of a pediatric hip specific outcome measure.

DETAILED DESCRIPTION:
1. Purpose Perthes disease is a hip disorder most often affecting children with an onset between four and eight years of age. The treatment options range from non-operative to bracing to operative intervention. As the disease most often affects the head of the femur, there is the potential for long-term conditions due to the residual hip joint deformity, following resolution of Perthes disease, leading to early degenerative hip osteoarthritis and potential impact on hip function, quality of life, and morbidity. A valid and reliable means by which to assess function and outcome is essential to determine the most effective means of treatment. Previous research has used different methods in different subject groups, making comparisons of results very difficult. Both the long-term outcome and change over time of a patient with Perthes disease could be measured with a hip joint specific patient oriented outcome measure. Several such measures have been developed in adults; specifically the Western Ontario and McMaster Osteoarthritis Scale (WOMAC) hip score are used very often. Though these tools have been well studied and validated in adults, they have not been tested or used in pediatric populations. As they were developed and shown to be valid, reliable, and responsive in adults, these measures require rigourous testing in pediatric populations prior to their use.
2. Hypothesis There is no true global hypothesis for the study since it is a validation/reliability study. There are hypotheses for each type of validity being studied.

   For construct validity (using convergence), the hypothesis would be a priori hypothesis in this study related to convergent validity is that, assuming the WOMAC has construct validity in this population, then the hip specific outcome scores should be different for each Stulberg classification stage.

   For construct validity (using extreme groups), the hypothesis would be a priori hypothesis in this study is that, assuming the measures have adequate construct validity in this population, the group of subjects being followed for treatment of an upper extremity fracture should have significantly better function, as indicated by a low score on the WOMAC and , compared to those with Perthes disease, who should have higher scores indicating poorer function.

   For criterion validity, the hypothesis would be a priori hypothesis related to criterion validity in this study predicts that, assuming adequate concurrent validity of these measures in this population, there should be a negative correlation between the Activities Scale for Kids - Performance (ASK-p, an activity level outcome score) and the WOMAC. The reason for a negative correlation is that high scores on the generic measure indicate better function, whereas low scores on the hip specific measures indicate better function.
3. Research Method All subjects enrolled in the study will be given the initial set of questionnaires at the time of recruitment and asked to complete them at home, following the clinical follow-up visit, and return the questionnaires by mail using a self-addressed, stamped envelope which will be provided. All subjects will complete the WOMAC. Those with healed Perthes disease will also complete the ASK-p at the first visit to the clinic following consent into the study. Those in the comparison group with an upper extremity fracture will not complete the generic measure. This will comprise the initial time point of the study. Those subjects who do not complete all required questionnaires, at this time point, will be excluded from the study. Radiographs of the affected hip and pelvis will be obtained for each patient with healed Perthes disease at the time of the clinic visit, which would be obtained regardless of inclusion in the study in the course of standard clinical follow-up.

   Those subjects with Perthes disease will also complete the WOMAC and measure two weeks following the initial time point. The questionnaires will be mailed to the subjects and they will be asked to complete the questionnaires and return them in a self-addressed, stamped envelope which will be provided. This will comprise the follow-up time point of the study. A reminder notification will be mailed at four weeks and a telephone call reminder at six weeks following the initial time point if the second series of questionnaires has not been returned. Those who do not complete the second series of questionnaires will be excluded from the reliability component of the study but maintained in the validity phase, provided the initial questionnaires were completed. Those with an upper-extremity fracture will not complete any additional questionnaires following the initial time point. The Stulberg classification will be determined, as outlined, following the initial time point but prior to analysis of the data.
4. Statistical Analysis All statistical analysis will be performed by a blinded, independent analyst. All analyses, with the exception of the weighted kappa statistic which will be calculated manually, will be performed with the use of S-PLUS software (version 6.2, Lucent Technologies, Inc.). The distribution of all questionnaire data will be determined with the use of frequency histograms to allow for the use of appropriate statistical tests. All statistical tests will be performed with α=0.05. The reported values will be the mean and the corresponding 95% confidence interval. Where two groups are compared, the mean difference between the groups and the 95% confidence interval of the difference will be reported.

There have been no previous studies or data of the WOMAC in a pediatric population. Using values obtained in studies of adults may not provide a good estimate for a power analysis in this population since other outcome measures, which have been validated in adults, have been shown to lack validity in children and adolescents. However, in order to estimate the sample size required for the correlation between the ASK-p and the hip outcome measures the previously reported adult derived values were required. On the basis of a minimum correlation of 0.6, which would be considered adequate, with α=0.05 and 80 per cent power, a total of 40 children are required for the study. Since there is no available evidence with which to estimate the correlation between these outcome measures, a liberal sample size will be recruited. In a similar study, except that generic as opposed to joint specific, outcome measures were used, a sample size of 196 subjects was recruited. Young et al recruited 200 subjects for their study in which several psychometric properties of the ASK-p were determined. A total of 200 subjects will be recruited across all centers participating in this study. There will be 100 subjects with an upper extremity fracture and 100 with healed Perthes disease. This sample size was chosen, in part, on the basis of the maximum number of subjects with healed Perthes which would be feasible to recruit over the time horizon of the study, which will be six months. It is anticipated that a minimum of four centers will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between 5-19 years
* Healed Perthes disease. Healed Perthes disease will be defined radiographically, in the accepted fashion, by the appearance of normal bone density of the femoral head. The restriction of those with Perthes disease to only those with resolution of the disease will prevent heterogeneity of the clinical presentation and anticipated functional abilities which would occur by including those in the acute phases of the disease, thereby reducing potential bias.
* All participants will have to be able to complete the questionnaires in English and, for those with Perthes disease, be able to complete the questionnaires again two weeks following the initial completion.

Exclusion Criteria:

* Amongst those being followed at the orthopaedic clinic of a participating center with an upper extremity fracture, those with a history of a hip disorder will be excluded. The reason for this is that these subjects will compose a comparison group with normal hip function, consequently a history of hip disorder would bias this comparison.
* Those with Perthes disease who demonstrate acute phases of the disease will be excluded. Acute phases of the disease will be defined in the accepted fashion, by the radiographic presence of fragmentation or reossification of the femoral head.
* Those who do not provide consent for participation in the study will be excluded, as will those who either cannot complete the questionnaire in English or are unable to complete a second set of questionnaires at two weeks.
* Those with cognitive impairment, precluding completion of the questionnaires, will be excluded.
* All those with concomitant medical problems will be excluded due to possible confounding of the clinical outcome measures.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children and adolescents, between the ages of five and nineteen years, being followed at the Orthopaedic clinic of a participating center with a diagnosis of an upper extremity fracture or healed Perthes disease will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Difference in WOMAC questionnaire scores between the five Stulberg classification stages in the Perthes group | Baseline

SECONDARY OUTCOMES:
Difference in WOMAC questionnaire scores between baseline and 2 weeks | Baseline to two weeks
Difference in WOMAC questionnaire scores between the Perthes and control group | Baseline
Correlation between WOMAC questionnaire and ASK-P scores in the Perthes group | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, MBBS, MS(Ortho), MHSc, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young NL, Williams JI, Yoshida KK, Wright JG. Measurement properties of the activities scale for kids. J Clin Epidemiol. 2000 Feb;53(2):125-37. doi: 10.1016/s0895-4356(99)00113-4. PMID 10729684